CLINICAL TRIAL: NCT00002087
Title: Safety, Tolerance, Efficacy and Pharmacokinetics of Multiple Doses of sCD4-PE40 in the Treatment of HIV-Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 084A; Amend 022; P/3325/0002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-04

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: Alvircept sudotox

SUMMARY:
To investigate the safety and tolerance of an increasing number of infusions per week of alvircept sudotox ( sCD4-PE40; soluble CD4-Pseudomonas exotoxin ) at a fixed dose when administered to HIV-1-infected individuals. To investigate the effect of sCD4-PE40 on the following parameters: T lymphocyte subsets, plasma HIV RNA and cellular HIV proviral DNA in PBMC and CD4 cells, p24 levels, serum beta-2 microglobulin, and neopterin levels.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity confirmed by Western blot.
* CD4 count of 100 - 500 cells/mm3 on a morning draw within 3 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Concurrent neoplasms other than basal cell carcinoma of the skin, in situ carcinoma of the cervix, or nondisseminated Kaposi's sarcoma.
* Hemophilia or other clotting disorders.
* Major organ allograft.
* Significant cardiac, hepatic, renal, or CNS disease.

Prior Medication:

Excluded:

* Antiretroviral agents within 2 months prior to study entry.
* Known anti-HIV medication within 60 days prior to study entry.
* Prior immunomodulators (e.g., systemic steroids, interferons, or interleukins) or other chemotherapy.

Prior Treatment:

Excluded:

* Prior radiation therapy. Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Univ Med Ctr, Stanford, California, United States

REFERENCES:
- [Background] Davey RT Jr, Boenning CM, Herpin BR, Batts DH, Metcalf JA, Wathen L, Cox SR, Polis MA, Kovacs JA, Falloon J, et al. Use of recombinant soluble CD4 Pseudomonas exotoxin, a novel immunotoxin, for treatment of persons infected with human immunodeficiency virus. J Infect Dis. 1994 Nov;170(5):1180-8. doi: 10.1093/infdis/170.5.1180. PMID 7963711